CLINICAL TRIAL: NCT02518880
Title: Dynamics of Stroke Volume and Cardiac Output During Parabolic Flight, and Its Relationship to Intravascular Volume
Acronym: DYMCO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 09-178
Record Dates: First submitted 2015-08-06; First posted 2015-08-10 (Estimated); Last update posted 2015-08-10 (Estimated); Status verified 2015-08

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Plasma volume measurements (Other)
  Interventions: Other: Parabolic flight; Other: plasma volume measurements

INTERVENTIONS:
Other: Parabolic flight
Other: plasma volume measurements

SUMMARY:
To understand the cardiovascular reactions of the human body to changing conditions of gravity is an important aim of space science. In this context, cardiac output (CO) is a key value to estimate the human cardiovascular system.

The main objective of this experiment is to determine the effects of parabolic flight on intravascular volume, and how these changes modulate the complex haemodynamics induced by the parabolas.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers (men or women),
* aged from 18 to 55,
* affiliated to a Social Security system,
* who accept to take part in the study,
* who have given their written stated consent,
* who already participated in parabolic flights (even in the same campaign)
* All subjects will pass a medical examination similar to a standard aviation medical examination for private pilot aptitude. There will be no additional test performed for subject selection

Exclusion Criteria:

* person who took part in a previous biomedical research protocol, of which exclusion period is not terminated,
* pregnant women

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2010-03; Primary Completion 2012-02 (Actual)

PRIMARY OUTCOMES:
haemoglobin concentration | baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Umr Ucbn/Inserm U1075 Comete, Caen, Basse-Normandie, France